CLINICAL TRIAL: NCT03981627
Title: A Randomized, Single-centre, Double-blind, 2-period Cross-over Trial to Assess Safety and Efficacy of ADO09 Versus Insulin Aspart in Subjects With Type 1 Diabetes Mellitus
Brief Title: A Trial to Assess Safety and Efficacy of ADO09 Versus Insulin Aspart in Subjects With Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Adocia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CT038-ADO09
Record Dates: First submitted 2019-06-07; First posted 2019-06-11 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Aspart

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Co-formulation of insulin analog and pramlintide (ADO09) (Experimental): Subcutaneous injection of ADO09 formulation
  Interventions: Drug: ADO09 formulation
- NovoRapid® (Active Comparator): Subcutaneous injection of insulin aspart
  Interventions: Drug: NovoRapid®

INTERVENTIONS:
Drug: ADO09 formulation — Subcutaneous injection of ADO09 formulation
  Arms: Co-formulation of insulin analog and pramlintide (ADO09)
Drug: NovoRapid® — Subcutaneous injection of insulin aspart
  Arms: NovoRapid®

SUMMARY:
This is a randomized, double-blind, active-controlled, 2 period cross-over clinical trial in subjects with type 1 diabetes mellitus using a Multiple Daily Injection (MDI) regimen.

DETAILED DESCRIPTION:
After a screening visit, eligible subjects will enter a run-in period. Subjects will receive a Continuous Glucose Monitoring (CGM) system for glucose monitoring and control at the beginning of the run-in and for the whole duration of the study. Each eligible subject will then be randomly allocated to a sequence of the 2 treatments, i.e. multiple daily injections of ADO09 and insulin aspart during 2 dosing periods. At Day 1 a mixed meal test (MMT) will be conducted at breakfast and subjects will remain at the clinical site until day 3. At Day 3 subjects will leave the clinical site and continue the treatment with IMP for the next 3 weeks. On Day 23 subjects will come back for a MMT on Day 24.

This study is constituted of 2 parts. In the first part (Part A), only subjects with daily prandial insulin dose ≤ 40 U/day will be enrolled.

Following the completion of the part A, an extension part (Part B) will be conducted to particularly assess the safety and tolerability of higher daily doses of ADO09 in patients with insulin requirements ≥ 40 U/day.

The clinical conduct and procedures will not change for the Extension Part of the study.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent obtained before any trial-related activities.
* Type 1 diabetes mellitus (as diagnosed clinically) ≥ 12 months.
* Treated with insulin ≥ 12 months.
* Using a multiple dosing insulin therapy (MDI) with basal and bolus insulin.
* HbA1c ≤ 9.0%.
* Fasting negative C-peptide (≤ 0.30 nmol/L).
* Total daily prandial dose: ≤ 40U in the Part A and ≥ 40 U in the Part B

Exclusion Criteria:

* Known or suspected hypersensitivity to products used in the clinical trial
* Type 2 diabetes mellitus
* Previous participation in this trial. Participation is defined as randomized.
* Receipt of any medicinal product in clinical development within 3 months before randomization in this trial.
* Known slowing of gastric emptying, including gastroparesis, and or gastrointestinal surgery that in the opinion of the investigator might change gastrointestinal motility and food absorption.
* Presence of clinically significant acute gastrointestinal symptoms (e.g. nausea, vomiting, heartburn or diarrhoea), as judged by the Investigator.
* Intake of medication known to affect gastrointestinal motility, including but not limited to erythromycin, metoclopramide, cisapride, cholestyramine or colestipol within 4 weeks before screening.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2020-06-27 (Actual); Study Completion 2020-06-27 (Actual)

PRIMARY OUTCOMES:
ΔAUCPG(0-4h) | From 0 to 4 hours
  Incremental area under the plasma glucose concentration-time curve from 0-4 hours after start of breakfast, assessed by Super GL at day 24.

SECONDARY OUTCOMES:
Pharmacokinetics of pramlintide | From 0 to 4 hours
  Area under the pramlintide concentration-time curve
Pharmacokinetics of insulins | From 0 to 4 hours
  Area under the insulins concentration-time curve
Plasma glucose control as measured by CGM | Over 24 hours
  Time and percentage of time in Range (TiR) [70-180] mg/dL
Safety and tolerability (Adverse Events recording) | Up to 24 days
  Number of Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Grit Andersen, MD, Principal Investigator — Profil Institut für Stoffwechselforschung GmbH
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany

REFERENCES:
- [Derived] Andersen G, Eloy R, Famulla S, Heise T, Meiffren G, Seroussi C, Gaudier M, Megret C, Chan YP, Soula O, Riddle M. A co-formulation of pramlintide and insulin A21G (ADO09) improves postprandial glucose and short-term control of mean glucose, time in range, and body weight versus insulin aspart in adults with type 1 diabetes. Diabetes Obes Metab. 2023 May;25(5):1241-1248. doi: 10.1111/dom.14972. Epub 2023 Jan 31. PMID 36633505